CLINICAL TRIAL: NCT06856538
Title: Analgesic Efficacy of Ultrasound-Guided Rhomboid Intercostal Sub Serratus Plane Block Versus Serratus Anterior Plane Block With General Anesthesia in Thoracotomy
Brief Title: Rhomboid Intercostal Sub Serratus Plane Block Versus Serratus Anterior Plane Block in Thoractomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yasser S Mostafa, MD (Other)
Responsible Party: Sponsor-Investigator, Yasser S Mostafa, MD, Lecturer, Fayoum University Hospital
Organization: Fayoum University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: D404
Record Dates: First submitted 2025-02-19; First posted 2025-03-04 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Thoracic; Pain
Keywords: Rhomboid intercostal block; serratus anterior plane block; Thoracotomy
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Ultrasonography

STUDY DESIGN:
Intervention Model Description: After endotracheal intubation, just before the block, the patients were randomly allocated into two groups based on a computerized randomization table created by a researcher who was not involved in the study. The researcher assigned a random ID to each patient, and a blinded anesthesiologist used this ID while collecting the postoperative data in the surgical ward.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Care Provider, Outcomes Assessor) Apart from the anesthesiologists who performed the blocks, all patients, surgeons, and postoperative nurses remained blinded to randomization throughout the study period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group R (Experimental): A high- frequency linear ultrasound transducer will be placed longitudinally (in the sagittal plane) on the patient's back, just 2 cm medial to the medial scapular border. Then, the probe will be slightly rotated to obtain an oblique parasagittal plane. The following landmarks will be identified: the trapezius muscle, rhomboid major muscle, intercostal muscles, pleura, and lungs (from superficial to deep in order of appearance). The rhomboid major muscle will be distinguished at the level of the T6 and T7 vertebrae, below the trapezius muscle.
  Interventions: Drug: Bupivacain; Device: Ultrasound
- Group S (Active Comparator): * The patient will be positioned laterally, and routine skin disinfection and draping will be completed.
  * Investigators also will use a linear ultrasound probe (Philips clear vue350, Philips healthcare, Andover MAO1810, USA, Machine ID: 1385, Nile medical center, service@nilemed.net) for performing the block.
  * The fifth rib will be identified along the mid-axillary line to locate the deep serratus anterior muscle and the superficial latissimus dorsi muscle.
  * The needle will be inserted between the fifth and fourth ribs using a 22G (50 mm) puncture needle.
  Interventions: Drug: Bupivacain; Device: Ultrasound

INTERVENTIONS:
Drug: Bupivacain — After the location will be confirmed through hydrodissection of 1 ml on the plane between the rhomboid major and the underlying intercostal muscles after confirming a negative aspiration via a a 22-gauge short bevel sonovisible needle (Spinocan, B. Braun Melsungen AG, Germany) using an in-plane technique then 10 ml of bupivacaine (concentration 0.25%) will be injected. and its spread will be manifested by the hydrodissection and widening of the plane visualized by ultrasound.
  Other Names: Marcaine 0.25%
Device: Ultrasound — A linear US transducer (Phillips-Saronno Italy) was placed vertically 3 cm lateral to the midline to visualize back muscles: the trapezius above, the rhomboid major in the middle, and the erector-spinae muscle on the bottom, as well as the TPs with shimmering pleura in between.

SUMMARY:
The objective of the current study is to compare the efficacy of the analgesic effect of ultrasound-guided unilateral Rhomboid intercostal and sub serratus plane block (RISS) versus Serratus anterior plane block (SAPB) in Thoracotomy incision.

DETAILED DESCRIPTION:
Open thoracotomy is commonly considered to be one of the most agonizing surgical operations. Pain following thoracotomy greatly impedes patient recovery and postoperative respiration. The pain experienced after a thoracotomy can originate from various factors, including the surgical incision, injury to the ribs and intercostal nerves, manipulation of the pleura and lung tissue, and the placement of a drainage tube.Recent advances in regional anesthesia techniques have aimed to provide more targeted and effective pain relief. Among these, ultrasound-guided fascial plane blocks, such as the rhomboid intercostal sub-serratus plane (RISS) block and the serratus anterior plane (SAP) block, have emerged as promising options. Both blocks target the thoracic nerves, but they differ in their anatomical approach and potential analgesic effects Postoperative pain was not only related to a comfortable recovery but also related to postoperative complications including pulmonary dysfunction, so the management of postoperative pain is an important part of the care of post operation.

Regional anesthesia techniques have been shown to have a good effect on postoperative analgesia and helps patients gain early recovery after operation.

Serratus anterior plane block (SAPB) is an easy, and safe method used for blockade of the sensory plane of the lateral cutaneous branch of the intercostal nerve (T2-T9).

The Serratus anterior plane block targets the lateral cutaneous branches of the thoracic intercostal nerves, which arise from the anterior rami of the thoracic spinal nerves and run in a neurovascular bundle immediately inferior to each rib. At the midaxillary line, the lateral cutaneous branches of the thoracic intercostal nerve traverse through the internal intercostal, external intercostal, and serratus anterior muscles innervating the musculature of the lateral thorax. These branches of the intercostal nerves travel through the two potential spaces described above.

The "Rhomboid intercostal and sub serratus plane block" (RISS) is a relatively newer block technique whose efficacy was documented in patients undergoing thoracic surgeries.

The RISS plane block involves the injection of local anesthetics into fascial planes, theoretically allowing for catheter placement to achieve continuous analgesia. Successful RISS plane blocks have been reported in various procedures, including lung transplantation, radical mastectomy, and nephrectomy, strongly suggesting favorable outcomes in postoperative pain relief.

In 2016, Elsharkawy et al. introduced a RA technique known as the rhomboid intercostal block (RIB). Rhomboid intercostal block involves injecting a local anesthetic into the upper intercostal muscle plane beneath the rhomboid muscles, providing analgesia to both the anterior and posterior thorax.Based on past studies, investigators found that RISS and SAPB are effectively decrease total opioid consumption, so investigators hypothesized one of them is the best.

Statistical analysis:

Statistical analysis will be conducted using IBM SPSS Statistics 22(IBM Corp., Armonk, NY, USA). The normal distribution of data will be assessed by the Kolmogorov-Smirnov and Shapiro-Wilk tests. Mean and standard deviation will be used as descriptive statistics for normally distributed numerical variables, while median and interquartile range (25th to 75th percentiles) will be used as descriptive statistics for non-normally distributed numerical variables. In addition, Chi-square test or fisher exact test will be employed to test the significance between categorical variables as appropriate. Independent t test will be employed for numerical data that exhibited normal distribution, whereas the Mann-Whitney test will be used for numerical data that did not adhere to normal distribution. A significance level of p < 0.05 will be deemed to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 years.
* Patients scheduled for unilateral Thoracotomy.
* American Society of Anesthesiologists (ASA) physical status I-III.
* Patients who are candidates for general anesthesia.
* No history of severe allergies to local anesthetics or other medications used during the procedure.

Exclusion Criteria:

* ASA PS class ≥ IV patients.
* obese (BMI ≥ 35) patients.
* Patients with uncontrolled cardiovascular.
* patients with neurological deficits, cardiopulmonary, hepatorenal , or metabolic diseases; anticoagulants; any drug allergies.
* Patients with emergency surgeries or re-do surgeries.
* Systemic infections or infections at the site of injection.
* Psychiatric illnesses (schizophrenia, bipolar, uncontrolled anxiety or depression).
* Narcotic dependency.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Total opioid consumption | 24 hours postoperatively.
  in microgram

SECONDARY OUTCOMES:
Total intraoperative opioid consumption | from begining of operation till 5 minutes after extubation
  in microgram
Visual analog pain score at rest | Immediately after the procedures
  Ranging from 0 indicating no pain to 10 indicating extreme pain
Visual analog pain score at cough | Immediately after the procedures
  Ranging from 0 indicating no pain to 10 indicating extreme pain
Visual analog pain score at rest | 1 hour postoperatively.
  Ranging from 0 indicating no pain to 10 indicating extreme pain
Visual analog pain score at cough | 1 hour postoperatively.
  Ranging from 0 indicating no pain to 10 indicating extreme pain
Visual analog pain score at rest | 3 hours postoperatively.
  Ranging from 0 indicating no pain to 10 indicating extreme pain
Visual analog pain score at cough | 3 hours postoperatively.
  Ranging from 0 indicating no pain to 10 indicating extreme pain
Visual analog pain score at rest | 6 hours postoperatively.
  Ranging from 0 indicating no pain to 10 indicating extreme pain
Visual analog pain score at cough | 6 hours postoperatively.
  Ranging from 0 indicating no pain to 10 indicating extreme pain
Visual analog pain score at rest | 12 hours postoperatively.
  Ranging from 0 indicating no pain to 10 indicating extreme pain
Visual analog pain score at cough | 12 hours postoperatively.
  Ranging from 0 indicating no pain to 10 indicating extreme pain
Visual analog pain score at rest | 24 hours postoperatively.
  Ranging from 0 indicating no pain to 10 indicating extreme pain
Visual analog pain score at cough | 24 hours postoperatively.
  Ranging from 0 indicating no pain to 10 indicating extreme pain
Time of first rescue analgesic | 5 minutes before first analgesic request
  in minutes
Baseline Heart rate | 5 minutes before anesthesia
  Beat / minute
Intraoperative Heart rate | every 30 minutes along operation
  Beat / minute
Baseline mean arterial blood pressure | 5 minutes before anesthesia
  mmHg
Intraoperative mean arterial blood pressure | every 30 minutes along operation
  mmHg
Baseline oxygen saturation | 5 minutes before anesthesia
  percentage with pulse oximetry
Intraoperative oxygen saturation | every 30 minutes along operation
  percentage with pulse oximetry
Total length of stay in hospital | 1-2 days
  in days
Patient satisfaction score | 12 hours after end of operation and extubation
  5 degree Likeart scale where 1 Extremely satisfied to 5 Extremely not satisfied
Incidence of hematoma | 30 minutes after nerve block
  Yes or no
Incidence of local anesthetic toxicity | 30 minutes after nerve block
  Yes or no
Incidence of nausea | 24 hours postoperative
  Yes or no
Incidence of vomiting | 24 hours postoperative
  Yes or no
Ramsay sedation score | 24 hours postoperative
  From 1 to 5 (1 Awake; agitated or restless or both - 2 Awake; cooperative, oriented, and tranquil - 3 Awake but responds to commands only - 4 Asleep; brisk response to light glabellar tap or loud auditory stimulus - 5 Asleep; sluggish response to light glabellar tap or loud auditory stimulus)
  Asleep; no response to glabellar tap or loud auditory stimulus

OTHER OUTCOMES:
Age | 5 minutes before entering operation department
  in years
Sex | 5 minutes before entering operation department
  Male of female

CONTACTS AND LOCATIONS:
Overall Officials: Mahdy A Abdelhady, MD, Study Chair — Fayoum University; Mohamed A Hamed, MD, Principal Investigator — Fayoum University; Mina M Sobhy, MD, Study Director — Fayoum University
Locations (1):
- Fayoum University hospital, El Fayoum Qesm, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altiparmak B, Korkmaz Toker M, Uysal AI, Dere O, Ugur B. Evaluation of ultrasound-guided rhomboid intercostal nerve block for postoperative analgesia in breast cancer surgery: a prospective, randomized controlled trial. Reg Anesth Pain Med. 2020 Apr;45(4):277-282. doi: 10.1136/rapm-2019-101114. Epub 2020 Feb 19. PMID 32079739
- [Background] Longo F, Piliego C. Rhomboid intercostal and subserratus plane block for non-intubated video-assisted thoracoscopic surgery. J Clin Anesth. 2020 May;61:109612. doi: 10.1016/j.jclinane.2019.09.006. Epub 2019 Oct 24. No abstract available. PMID 31668692
- [Background] Hassan ME, Wadod MAA. Serratus anterior plane block and erector spinae plane block in postoperative analgesia in thoracotomy: A randomised controlled study. Indian J Anaesth. 2022 Feb;66(2):119-125. doi: 10.4103/ija.ija_257_21. Epub 2022 Feb 24. PMID 35359482